CLINICAL TRIAL: NCT01438788
Title: Low Protein Diet to Correct Defective Autophagy in Patients With Collagen VI Related Myopathies
Brief Title: Low Protein Diet in Patients With Collagen VI Related Myopathies
Acronym: LPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOR-0018156
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Bethlem Myopathy; Ullrich Congenital Muscular Dystrophy
Keywords: Bethlem myopathy; Ullrich congenital muscular dystrophy; Low protein diet; Autophagy; Pilot clinical trial
MeSH Terms: conditions — Bethlem myopathy; Scleroatonic muscular dystrophy | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients on a low protein diet (Experimental)
  Interventions: Other: Low protein diet

INTERVENTIONS:
Other: Low protein diet — Patients will receive a diet with 0.6-0.8 grams of protein/kilogram body weight/day for one year. Bread, biscuits and pasta will be in part substituted with aproteic food.

SUMMARY:
* This is a 2 stage exploratory study with a 3-month observational phase on the natural course, followed by a 12-month, open-label, non-comparative, single-arm, phase II pilot study on the efficacy, safety and tolerability of a low-protein diet (LPD) in 8 adult patients with Bethlem myopathy (BM) and Ullrich congenital muscular dystrophy (UCMD).
* Objective of this trial is to test the effect of a normocaloric LPD to reactivate autophagy in BM/UCMD patients. The primary end point of the study will be the change in muscle biopsy of Beclin 1, a marker of autophagy, at 1 year of LPD treatment when compared to baseline.
* The rationale rests on our discoveries that (i) mitochondrial dysfunction mediated by inappropriate opening of the PTP plays a key role in collagen VI myopathies; (ii) defective autophagy with impaired removal of defective mitochondria amplifies the defect; and (iii) reactivation of autophagy with a low-protein diet or treatment with cyclosporine A, the mitochondrial PTP inhibitor, cured Co6a1-/- mice, hinting at a common target among all beneficial treatments - namely autophagy.
* Specific aims of this project are to (i) study the modifications of clinical, nutritional and laboratory parameters in a cohort of patients with BM/UCMD during a 3-month observational period before starting the LPD treatment; (ii) assess the effect of a normocaloric LPD in correcting defective autophagy in muscle of patients; (iii) test if new non-invasive biomarkers of activation of autophagy examined in the blood are mirroring the effect of LPD in the muscle biopsy; (iv) assess the clinical efficacy and safety of the LPD with an innovative combination of complementary measures of the nutritional status in patients.
* The anticipated output is defining and validating a therapeutic nutritional approach in autophagy upregulation for BM/UCMD.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years.
* Women of childbearing age must have a negative pregnancy test and must use adequate contraception during the study.
* Clinical and molecular diagnosis of Bethlem myopathy or Ullrich congenital muscular dystrophy.
* No previous treatment with CsA within 6 months prior to the start of the study.
* Willing and able to adhere to the study visit schedule and other protocol requirements.
* Written informed consent signed.

Exclusion Criteria:

* Current or history of liver or renal disease.
* Pregnant or breast-feeding women.
* Any serious internal medicine condition interfering with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Reactivation of autophagy measured as a change in Beclin 1 as a marker of autophagy in muscle biopsy from baseline (Day 1) to Day 365 | one year

SECONDARY OUTCOMES:
Assess the safety of a LPD in patients with BM/UCMD . Nutritional parameters . Muscle mass . Muscle strength | one year

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Merlini, MD, Principal Investigator — Istituto Ortopedico Rizzoli, Bologna, Italy
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Grumati P, Coletto L, Sabatelli P, Cescon M, Angelin A, Bertaggia E, Blaauw B, Urciuolo A, Tiepolo T, Merlini L, Maraldi NM, Bernardi P, Sandri M, Bonaldo P. Autophagy is defective in collagen VI muscular dystrophies, and its reactivation rescues myofiber degeneration. Nat Med. 2010 Nov;16(11):1313-20. doi: 10.1038/nm.2247. Epub 2010 Oct 31. PMID 21037586
- [Result] Castagnaro S, Pellegrini C, Pellegrini M, Chrisam M, Sabatelli P, Toni S, Grumati P, Ripamonti C, Pratelli L, Maraldi NM, Cocchi D, Righi V, Faldini C, Sandri M, Bonaldo P, Merlini L. Autophagy activation in COL6 myopathic patients by a low-protein-diet pilot trial. Autophagy. 2016 Dec;12(12):2484-2495. doi: 10.1080/15548627.2016.1231279. Epub 2016 Sep 22. PMID 27656840